CLINICAL TRIAL: NCT02836470
Title: A Randomized, Double-Blind, Placebo-Controlled Proof of Concept Study to Evaluate LB1148 for Return of Gastrointestinal Function, Post-Operative Ileus and Intra-Abdominal Adhesions in Subjects Undergoing Elective Bowel Resection
Brief Title: A Study to Evaluate LB1148 for Return of Gastrointestinal Function and Adhesions in Subjects Undergoing Bowel Resection
Acronym: PROFILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palisade Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBS-POI-201
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-04

CONDITIONS: Ileus; Post-Operative Adhesions
Keywords: Post-operative Ileus; Post-Operative Abdominal Adhesions; Return of Gastrointestinal Function; Anastomosis; Enterotomy; Enterostomy; Colorectal Surgery; Intestines Surgery
MeSH Terms: conditions — Ileus | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LB1148 (Experimental): Active
  Interventions: Drug: LB1148
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LB1148 — A total of 700 mL of drug product will be administered orally as a split dose before surgery.
  Other Names: Active
  Arms: LB1148
Drug: Placebo — A total of 700 mL of placebo will be administered orally as a split dose before surgery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish preliminary evidence of the efficacy, safety, and tolerability of LB1148 for the treatment of post-operative ileus and intra-abdominal adhesions in subjects undergoing elective bowel resection.

DETAILED DESCRIPTION:
This will be a multicenter, randomized, double-blind, parallel, placebo-controlled, proof-of-concept, adaptive design, Phase 2 study to evaluate LB1148 for return of gastrointestinal function and reduction of post-operative ileus and intra-abdominal adhesions in subjects undergoing elective bowel resection surgery with or without a planned stoma.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for participation in the study only if they meet ALL of the following inclusion criteria:

1. Scheduled to undergo an elective (non-emergent) bowel resection with a planned stoma via laparotomy or minimally invasive technique. This includes any subject in which a resection of the small intestine, colon, or rectum is performed for any elected indication.
2. Planned stoma takedown or other planned abdominal surgery within 8 months of the initial surgery.
3. Willing to perform and comply with all study procedures including attending clinic visit as scheduled and completion of a second surgery for stoma takedown or other abdominal surgery and to determine the presence of intra-abdominal adhesions.
4. Has been informed of the nature of the study (either the subject or their legal representative), agrees to its provisions, and has provided written informed consent.

Exclusion Criteria:

Subjects will not be eligible for participation in the study if they meet ANY of the following exclusion criteria:

1. <18 or >80 years of age.
2. Requires emergency bowel surgery.
3. Has had 1 or more abdominal surgeries, excluding the current, for inflammatory bowel disease, including, but not limited to, inflammatory bowel disease (IBD), Crohn's Disease, or ulcerative colitis.

   Note: This does not apply to previous surgery such as hernia repair unrelated to IBD.
4. American Society of Anesthesiologists (ASA) Class 4 or 5.
5. Known inability to take the study drug orally (i.e. complete small bowel obstruction).
6. Has contraindications or potential risk factors to taking TXA. These include subjects with:

   1. Known sensitivity to TXA;
   2. Recent craniotomy (past 30 days);
   3. Active cerebrovascular bleed;
   4. Active thromboembolic disease (such as deep vein thrombosis, pulmonary embolism, cerebral thrombosis, ischemic stroke, or acute coronary syndrome);
   5. Acute promyelocytic leukemia taking all-trans retinoic acid for remission induction, or
   6. Continuing use of a combined hormonal contraceptive and or combined hormonal replacement therapy (including combined hormonal pill, patch, or vaginal ring).
7. Has peritoneal carcinomatosis
8. History of or current seizure disorder.
9. Patients with myeloproliferative disorders.
10. Any other condition that, in the opinion of the Investigator, would preclude the subject from being an appropriate candidate for the study, including severe renal or hepatic impairment.
11. Planned treatment with alvimopan (Entereg®) during study participation period.
12. Planned use of 4% icodextrin (Adept®) or SEPRAFILM during the first surgery.
13. Received any other investigational therapy within 4 weeks prior to Randomization
14. Female subjects of childbearing potential with a positive urine or serum pregnancy test or who are not taking (or not willing to take) acceptable birth control measures (abstinence, intrauterine devices, contraceptive implants or barrier methods) through Day 30. Additionally, those women who are lactating and insist on breast feeding within 5 days of the last dose of study drug.
15. Known history of radiation enteritis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Jones, MD, Study Director — CMO
Locations (28):
- United States (28):
  - Site 315, Mobile, Alabama
  - Site 307, Yuma, Arizona
  - Site 329, Irvine, California
  - Site 310, Pasadena, California
  - Site 302, Sylmar, California
  - Site 312, Torrance, California
  - Site 306, Clearwater, Florida
  - Site 303, Miami, Florida
  - Site 331, Miami, Florida
  - Site 305, Miami, Florida
  - Site 308, Orlando, Florida
  - Site 328, Louisville, Kentucky
  - Site 321, Baltimore, Maryland
  - Site 324, Burlington, Massachusetts
  - Site 325, Rochester, Minnesota
  - Site 317, New York, New York
  - Site 323, New York, New York
  - Site 318, Chapel Hill, North Carolina
  - Site 301, Cleveland, Ohio
  - Site 322, Pittsburgh, Pennsylvania
  - Site 330, Wynnewood, Pennsylvania
  - Site 327, Charleston, South Carolina
  - Site 320, Dallas, Texas
  - Site 316, Fort Worth, Texas
  - Site 311, Houston, Texas
  - Site 319, Houston, Texas
  - Sie 309, Houston, Texas
  - Site 326, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LB1148: Active
  LB1148: A total of 700 mL of drug product was administered orally as a split dose before surgery.
- Placebo: Placebo
  Placebo: A total of 700 mL of placebo was administered orally as a split dose before surgery.
Period: Overall Study
Arm/Group | LB1148 | Placebo
Started | 57 | 55
Completed | 52 | 49
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LB1148 | Placebo | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (11.56) | 55.9 (13.94) | 57.6 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 33 | 31 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 52 | 49 | 101
  Black | 3 | 3 | 6
  Asian | 0 | 1 | 1
  American Indian | 0 | 0 | 0
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 57 | 55 | 112

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Extent and Severity of Intra-abdominal Adhesions Among Subjects Treated With LB1148 or Placebo
Description: Extent and severity of intra-abd. adhesions will be determined by the surgeon using the "Intra-Abdominal Adhesion Extent and Severity Assessment Worksheet" with a min. value of zero (0) (better) and a max. value of one hundred and eight (108) (worse). And which records four (4) Sub scores for nine (9) abd. regions which are all summed to make the Total Extent and severity score. Sub scores include: 1) Abd. Wall to Bowel Extent Score (0-3); 2) Abd. Wall to Bowl Severity Score (0-3); Bowel to Bowel (or Viscera) Extent Score (0-3); Bowel to Bowel (or Viscera) Severity Score (0-3); The nine (9) Abd. Regions include: Right upper; Epigastrium; Left upper; Left flank; Left lower; Pelvis; Right lower; Right flank; and Central. Each Sub score is scored with a min. value of zero (0) (better) and a max. value of three (3) (worse); 0=no adhesion; 1=min. (<1/3 of the site is covered); 2=mod. (1/3 to 2/3 of the site is covered); 3=extensive (>2/3 of the site is covered).
Time Frame: up to 8 months from the index surgery
Population: The protocol from July 11 '16 underwent 6 amendments. The Safety Population included all randomized subjects (n=112). The modified Intention to Treat (mITT) population comprised subjects meeting criteria and receiving full dose with no key deviations (n=33). Those completing per protocol (PP) were (n=22). The smaller evaluable populations for Outcome Measures vs. Safety Population are due to Second Surgery completion requirements.
Measure: Mean (Standard Deviation); unit: total extent and severity scores
Arm/Group | LB1148 | Placebo
Number analyzed (Participants) | 11 | 11
total extent and severity scores
  Minimally Invasive Approach: number analyzed (Participants) | 10 | 9
  Minimally Invasive Approach | 20.3 (23.77) | 4.3 (5.87)
  Laparotomy Approach: number analyzed (Participants) | 1 | 2
  Laparotomy Approach | 4.0 (NA) — not applicable as there was only 1 subject (LB1148) in this group | 8.5 (9.19)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from first administration of study drug through initial hospital discharge, or early termination, whichever came first. Following discharge through the second surgery visit, if applicable, any hospital readmissions were collected. Any serious adverse event or adverse event related to the second surgery was also collected from Day 0 to Month 3 ±1 Month.
Arm/Group | LB1148 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/57 | 0/55
Serious Adverse Events (participants affected / at risk) | 16/57 | 14/55
Other Adverse Events (participants affected / at risk) | 38/57 | 40/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LB1148 (N=57) | Placebo (N=55)
Post operative ileus (Injury, poisoning and procedural complications) | 2 | 6
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
anal fissure (Gastrointestinal disorders) | 1 | 0
gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
chest pain (General disorders) | 1 | 0
pyrexia (General disorders) | 0 | 2
abdominal abscess (Infections and infestations) | 1 | 0
abdominal sepsis (Infections and infestations) | 0 | 1
pelvic abscess (Infections and infestations) | 1 | 0
peritonitis (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 1 | 0
sepsis (Infections and infestations) | 0 | 2
septic shock (Infections and infestations) | 0 | 1
vascular device infection (Infections and infestations) | 1 | 0
wound infection (Infections and infestations) | 0 | 1
anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
procedural pain (Injury, poisoning and procedural complications) | 1 | 0
splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
dehydration (Metabolism and nutrition disorders) | 0 | 1
acute kidney injury (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
urinary retention (Renal and urinary disorders) | 1 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1
acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LB1148 (N=57) | Placebo (N=55)
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Urinary retention (Renal and urinary disorders) | 5 | 1
anemia (Blood and lymphatic system disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6
Pneumonia (Infections and infestations) | 3 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 4 | 8
Procedural pain (Injury, poisoning and procedural complications) | 6 | 4
nausea (Gastrointestinal disorders) | 12 | 12
pyrexia (General disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT02836470/Prot_002.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT02836470/SAP_003.pdf